CLINICAL TRIAL: NCT07169201
Title: A High-Temporal Resolution CT Platform for Imaging and Functional Evaluation of Heart
Brief Title: High-Resolution CT for Heart
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HiTe-CT
Record Dates: First submitted 2025-08-02; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort for CT-RWS: This cohort includes patients with suspected or known coronary artery disease undergoing coronary CTA using a high-temporal-resolution CT scanner (uCT SiriuX Pro). Patients must have at least one lesion with moderate-to-severe stenosis (≥50%) on CTA. All participants will subsequently undergo invasive coronary angiography and OCT. The study aims to assess the correlation between CT-derived radial wall strain (CT-RWS) and OCT-defined plaque vulnerability features, including thin-cap fibroatheroma (TCFA), lipidic plaque burden, and lipid-to-cap ratio (LCR). CT-RWS will be derived from coronary CTA using a dedicated algorithm. OCT will serve as the invasive reference for plaque characterization. No investigational drug or device will be used. Lesion-level comparisons will evaluate whether CT-RWS can serve as a non-invasive surrogate of plaque biomechanics.
  Interventions: Diagnostic Test: Angiography based RWS and OCT based plaque characteristcis
- Cohort for myocardial bridging: This cohort includes patients with myocardial bridging (MB) identified on coronary CTA using a high-temporal-resolution CT scanner (uCT SiriuX Pro). Patients must have symptoms suggestive of ischemia and elevated systolic flow perfusion ratio (CT-SFPR), a novel CT-based index designed to quantify dynamic systolic compression of the bridged coronary segment. Eligible patients will undergo invasive coronary angiography with physiological assessment using resting full-cycle ratio (RFR) to evaluate the functional significance of MB. The primary objective is to assess the correlation between CT-SFPR and invasively measured RFR. CT-SFPR will be calculated from multiphase coronary CTA using a dedicated post-processing algorithm. No investigational drugs or devices are involved. The cohort aims to validate CT-SFPR as a non-invasive marker for MB-related ischemia.
- Cohort for prognosis: This cohort includes patients with suspected or known coronary artery disease who undergo coronary CTA using a high-temporal-resolution CT scanner (uCT SiriuX Pro). CT-derived radial wall strain (CT-RWS) will be calculated for coronary lesions using a dedicated post-processing algorithm. All patients will be followed prospectively for up to 2 years to monitor the occurrence of major adverse cardiovascular events (MACE), including cardiac death, non-fatal myocardial infarction, and target vessel revascularization. The primary objective is to assess the prognostic value of CT-RWS for predicting future cardiovascular events. CT-RWS will be analyzed both as a continuous variable and based on predefined thresholds to identify high-risk plaque biomechanics. No investigational interventions will be applied. This cohort aims to validate CT-RWS as a non-invasive imaging biomarker for long-term risk stratification.

INTERVENTIONS:
Diagnostic Test: Angiography based RWS and OCT based plaque characteristcis — Angiography based RWS and OCT based plaque characteristcis
  Groups: Cohort for CT-RWS

SUMMARY:
This prospective observational study aims to evaluate a high-resolution coronary CT platform (uCT SiriuX Pro) for non-invasive assessment of coronary plaque biomechanics and functional physiology in high-risk patients. The system enables CT-derived radial wall strain (CT-RWS), a novel biomarker reflecting plaque vulnerability, with potential correlation to invasive OCT findings and clinical outcomes.

The study will assess the diagnostic performance and prognostic value of CT-RWS, along with a new CT-based index of systolic flow perfusion (CT-SFPR) for evaluating the hemodynamic relevance of myocardial bridging, compared to nuclear perfusion imaging. Additionally, left ventricular ejection fraction derived from dynamic CTA (CT-EF) will be compared with echocardiography to evaluate its feasibility and accuracy. This is the first study to comprehensively validate CT-RWS, CT-SFPR, and CT-EF using a fully non-invasive, high-temporal-resolution CT platform.

DETAILED DESCRIPTION:
Vulnerable coronary plaques remain a major cause of adverse cardiac events, including myocardial infarction and cardiac death, even in lesions that are not flow-limiting by conventional assessment. Invasive imaging modalities such as optical coherence tomography (OCT) have enabled identification of high-risk plaque features, including thin-cap fibroatheroma (TCFA), large lipid pools, and high lipid-to-cap ratio (LCR), which are linked to plaque rupture and clinical instability. However, the widespread use of OCT is limited by cost, technical demands, and the need for invasive catheterization.

Radial wall strain (RWS) has emerged as a novel imaging biomarker reflecting local plaque biomechanics. Studies based on angiography-derived RWS, such as those by Wang et al. (JACC Cardiovasc Interv 2025) and Hong et al. (EuroIntervention 2023), have shown that high RWS is significantly associated with OCT-defined vulnerable plaque features and predictive of future cardiovascular events, particularly in high-risk populations. Despite this promise, angiographic RWS still requires invasive procedures.

To overcome this limitation, the investigators have developed a non-invasive imaging platform: the uCT SiriuX Pro, an advanced cardiac CT scanner designed by United Imaging Healthcare. With a leading gantry rotation speed of 0.229 seconds, this system enables ultra-high temporal resolution, supporting high-fidelity cardiac cine imaging, spectral imaging, and integrated perfusion-angiography acquisition. These capabilities allow for the first-time derivation of CT-based radial wall strain (CT-RWS) from coronary CT angiography (CTA), offering a novel, fully non-invasive surrogate for assessing plaque biomechanics. This technology has not been previously documented in the literature.

In addition to evaluating plaque vulnerability, the study also aims to assess myocardial bridging (MB), a congenital anomaly often regarded as benign but increasingly linked to ischemia and adverse outcomes. Using high-temporal-resolution CT, the investigators propose to derive a new index-the systolic flow perfusion ratio (CT-SFPR)-to quantify dynamic coronary compression and its hemodynamic impact. The diagnostic relevance of CT-SFPR will be compared with established perfusion deficits identified on nuclear imaging.

Furthermore, the advanced temporal resolution of uCT SiriuX Pro enables dynamic volumetric analysis of left ventricular function. This study will also evaluate CTA-derived ejection fraction (CT-EF) in comparison with echocardiography to validate its feasibility and accuracy for non-invasive cardiac function assessment.

This prospective observational registry will enroll high-risk patients with suspected or known coronary artery disease. It aims to systematically validate CT-RWS, CT-SFPR, and CT-EF against invasive and functional imaging benchmarks and to assess their prognostic significance during clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years with suspected or known CAD or with type 2 diabetes

Exclusion Criteria:

* those can not undergo CTA and angiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, we consecutively enrolled patients who were either suspected or diagnosed with coronary artery disease (CAD) in the outpatient setting, as well as those with diabetes presenting with atypical symptoms. Patients were eligible for inclusion if they were willing to undergo coronary CT angiography (CTA) followed by invasive coronary angiography. Major exclusion criteria included contrast agent allergy, impaired renal function, a history of coronary artery bypass grafting, and any other condition deemed unsuitable for CTA or invasive coronary angiography.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
correlation between CT-RWS and Angiography-derived RWS/OCT-detected vulnerable plaque features | Perioperative/Periprocedural
  We will measure the RWS derived from coronary CT angiography (CT-RWS). After patients undergo coronary angiography and OCT examinations, we will also measure the angiography-derived RWS, both expressed as percentages. Correlation analyses will be performed to investigate the association between CT-RWS and angiography-derived RWS. In addition, OCT plaque characteristics, including thin-cap fibroatheroma, lipidic plaque burden, and lipid-to-cap ratio, will be assessed. Correlation analyses will be conducted to explore the relationships between CT-RWS and these OCT-derived plaque characteristics.

SECONDARY OUTCOMES:
CT perfsusion and myocardial bridging | Baseline
  To evaluate a novel CT-derived Systolic Flow Perfusion Ratio (CT-SFPR) for myocardial bridging lesions, by comparison with ischemia detected on SPECT.

OTHER OUTCOMES:
prognostic value of CT-RWS | from enrollment to 3-year follow up
  To assess the prognostic value of CT-RWS for major adverse cardiovascular events (MACE) during 3-year follow-up.